CLINICAL TRIAL: NCT07070479
Title: A Bayesian Adaptive Phase II Randomized Trial Comparing Ivonescimab, Ivonescimab Plus Nimotuzumab, Liposomal Mitoxantrone Plus Anti-PD-1 Antibody, and Liposomal Irinotecan Plus S-1 in Patients With PD-1-Resistant Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Combination Therapy for PD-1 Resistant Recurrent or Metastatic Nasopharyngeal Carcinoma: A Bayesian Adaptive Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.BYAFZZX.034
Record Dates: First submitted 2025-06-24; First posted 2025-07-17 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; Recurrent; metastatic; PD-1 resistance; Bayesian adaptive design; Ivonescimab; Nimotuzumab; Liposomal mitoxantrone; Liposomal irinotecan; S-1
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — nimotuzumab; irinotecan sucrosofate; S 1 (combination); Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ivonescimab Monotherapy (Experimental): Participants will receive Ivonescimab at a dose of 10 mg/kg via intravenous infusion, Q3W. Treatment will continue until the occurrence of intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, loss to follow-up, or death, whichever occurs first.
  Interventions: Drug: Ivonescimab
- Ivonescimab plus Nimotuzumab (Experimental): Participants will receive Ivonescimab at a dose of 10 mg/kg via intravenous infusion, combined with Nimotuzumab 400 mg via intravenous infusion, Q3W.
  Treatment will continue until the occurrence of intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, loss to follow-up, or death, whichever occurs first.
  Interventions: Drug: Ivonescimab; Drug: Nimotuzumab
- Mitoxantrone Plus PD-1 Inhibitor (Experimental): Participants will receive mitoxantrone hydrochloride liposome at 20 mg/m² via intravenous infusion, combined with a PD-1 inhibitor - either tislelizumab (200 mg/cycle), camrelizumab (200 mg/cycle), or toripalimab (240 mg/cycle) - Q3W, for up to 8 cycles.
  After combination therapy, participants will continue receiving PD-1 blockade monotherapy every 3 weeks for up to 2 years, or until the occurrence of intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, loss to follow-up, or death, whichever occurs first.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome; Drug: PD-1 Inhibitors
- Irinotecan plus S-1 (Experimental): Participants will receive liposomal irinotecan at 50 mg/m² via intravenous infusion on D1 and D15, Q4W, in combination with oral S-1 administered BID on D 1-14 of each cycle, for up to 6 cycles.
  The dose of S-1 is based on body surface area (BSA). BSA < 1.25 m²: 40 mg per dose ; 1.25 m² ≤ BSA < 1.5 m²: 50 mg per dose; BSA ≥ 1.5 m²: 60 mg per dose Treatment will continue until the occurrence of intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, loss to follow-up, or death, whichever occurs first.
  Interventions: Drug: Irinotecan liposome; Drug: S-1

INTERVENTIONS:
Drug: Ivonescimab — Ivonescimab 10 mg/kg via intravenous infusion, until the occurrence of intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, loss to follow-up, or death, whichever occurs first.
  Arms: Ivonescimab Monotherapy; Ivonescimab plus Nimotuzumab
Drug: Nimotuzumab — Nimotuzumab 400 mg via intravenous infusion, Q3W, until the occurrence of intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, loss to follow-up, or death, whichever occurs first.
  Arms: Ivonescimab plus Nimotuzumab
Drug: Irinotecan liposome — Irinotecan liposome 50mg/m2 via intravenous infusion, D1, D15, Q4W for up to 6 cycles or until intolerable toxicity, subject withdrawal of informed consent, diseases progression, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first.
  Arms: Irinotecan plus S-1
Drug: S-1 — S-1, D1-D14, BID, p.o., (BSA < 1.25 m2, 40 mg/dose; 1.25 m2 ⩽ BSA < 1.5 m2, 50 mg/dose; BSA ⩾ 1.5 m2, 60mg/dose), Q4W for up to 6 cycles or until intolerable toxicity, subject withdrawal of informed consent, diseases progression, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first.
  Arms: Irinotecan plus S-1
Drug: Mitoxantrone Hydrochloride Liposome — Mitoxantrone hydrochloride liposome 20mg/m2 via intravenous infusion, Q3W for up to 8 cycles or until intolerable toxicity, subject withdrawal of informed consent, diseases progression, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first
  Arms: Mitoxantrone Plus PD-1 Inhibitor
Drug: PD-1 Inhibitors — PD-1 blockade (comprising tislelizumab <200 mg/cycle>, carrellimab <200 mg/cycle>, or toripalimab <240 mg/cycle>) , Q3W for two years, or until intolerable toxicity, subject withdrawal of informed consent, diseases progression, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first.
  Arms: Mitoxantrone Plus PD-1 Inhibitor

SUMMARY:
This is a prospective, Bayesian adaptive, phase II clinical trial designed to evaluate the safety and efficacy of four treatment regimens in patients with recurrent (unamenable to local therapy) or metastatic nasopharyngeal carcinoma (NPC) who have failed after at least one prior platinum-containing standard regimen and anti-PD-1/PD-L1 therapy.

The four treatment arms include:

1. Ivonescimab monotherapy,
2. Ivonescimab combined with nimotuzumab,
3. Liposomal mitoxantrone plus anti-PD-1 antibody, and
4. Liposomal irinotecan plus S-1.

DETAILED DESCRIPTION:
Patients with recurrent (not amenable to local therapy) or metastatic nasopharyngeal carcinoma (NPC) who have progressed after at least one prior platinum-containing standard regimen and anti-PD-1/PD-L1 therapy are eligible for this study. This trial adopts a Bayesian Adaptive Randomization with Constant Power parameter (BARCP) design. The planned maximum sample size is 208 patients, with a minimum of 32 patients to be enrolled before potential early termination for futility or efficacy based on interim analysis.

The first 40 patients will be randomized with equal probability to one of the four treatment arms:

1. Ivonescimab monotherapy
2. Ivonescimab combined with nimotuzumab
3. Liposomal mitoxantrone plus an anti-PD-1 antibody
4. Liposomal irinotecan plus S-1

Subsequent randomization probabilities will be updated based on objective response rate (ORR) using interim analyses, which will include decisions for early efficacy, futility, or reassignment of allocation probabilities for future participants. Interim analyses will be conducted every time 16 new patients complete ORR assessment. The minimum allocation probability for each treatment arm is constrained to 5%.

All patients will receive treatment until disease progression (as determined by the investigator based on RECIST 1.1 criteria), intolerable toxicity, withdrawal of informed consent, initiation of new anticancer therapy, loss to follow-up, death, or study completion-whichever occurs first. Regular visits and imaging assessments will be conducted to evaluate the efficacy and safety of the treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed recurrent or metastatic non-keratinizing nasopharyngeal carcinoma (either differentiated or undifferentiated subtype, corresponding to WHO type II or III).
2. Age between 18 and 70 years.
3. Performance Status (PS) score of 0 or 1.
4. Disease progression after prior platinum-based doublet chemotherapy.
5. Received at least one line of systemic therapy previously. (Progression occurring during or within 6 months after definitive concurrent chemoradiotherapy, neoadjuvant/adjuvant therapy, or treatment completion may be counted as first-line treatment.)
6. Resistance to anti-PD-1 antibody therapy (either combination or sequential), including primary or secondary resistance（PD-1 exposure must be at least 6 weeks.）
7. At least one measurable lesion according to RECIST 1.1 criteria.
8. All acute toxicities from prior anti-tumor therapies have resolved to grade ≤1 (per NCI-CTCAE v5.0) or meet the specified inclusion/exclusion thresholds. (Certain toxicities such as alopecia, hair color changes, nail changes, fatigue, etc., which do not pose safety risks, are exempt.)
9. Adequate organ function:

   Hematology: WBC ≥ 4000/μL, absolute neutrophil count ≥ 2000/μL, hemoglobin ≥ 9 g/dL, platelets ≥ 100,000/μL.

   Liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (patients with Gilbert's syndrome and bilirubin ≤ 3 × ULN are eligible); AST and ALT ≤ 3 × ULN; alkaline phosphatase ≤ 3 × ULN; albumin ≥ 3 g/dL.

   Coagulation: INR, prothrombin time (PT), or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.

   Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min calculated by Cockcroft-Gault formula. Proteinuria: Urine protein/creatinine ratio (UPC) < 1.0. For UPC ≤ 0.5, no further testing is required; for UPC > 0.5, 24-hour urine protein must be < 1000 mg for eligibility.
10. Estimated life expectancy of at least 3 months.
11. Signed informed consent and willingness and ability to comply with study visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Locoregional recurrent lesions that are amenable to definitive (curative) treatment, such as surgery.
2. Prior treatment with any regimen included in the study protocol.
3. Prior use of agents targeting the VEGF or VEGFR pathway.
4. Diagnosis and/or treatment of another malignancy within the past 5 years, with the exception of adequately treated carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ.
5. Receipt of surgery, chemotherapy, radiotherapy, immunotherapy, any investigational agent, or other anti-cancer therapy within 4 weeks prior to enrollment (or within 2 weeks for palliative radiotherapy).
6. Tumor encasement of the internal carotid artery or evidence of nasopharyngeal necrosis observed on endoscopy prior to enrollment.
7. Any significant bleeding event (≥ Grade 2, CTCAE v5.0) within 4 weeks prior to enrollment, or visible hemoptysis defined as ≥ 1/2 teaspoon of fresh red blood or blood clots with little or no sputum. Recurrent positive fecal occult blood test (++ or more) during screening also leads to exclusion. (Patients with occasional blood-tinged sputum may be eligible.)
8. Active peptic ulcers or gastrointestinal surgery within 1 month prior to enrollment; history within 6 months of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, gastrointestinal hemorrhage, esophageal varices, or pathological fracture.
9. Uncontrolled hypertension (systolic >140 mmHg or diastolic >90 mmHg) despite antihypertensive therapy; coronary artery disease ≥ Grade II; or any of the following within 6 months prior to enrollment: myocardial infarction, severe or unstable angina, NYHA class II or higher heart failure, sustained arrhythmia ≥ Grade 2 (including QTc >450 ms in males or >470 ms in females), atrial fibrillation of any grade, coronary or peripheral artery bypass grafting, symptomatic congestive heart failure, or cerebrovascular events (e.g., TIA or symptomatic pulmonary embolism). History of arterial thromboembolism or venous thromboembolism > Grade 3. (ST elevation ≥2 mm on ECG without clinical evidence of myocardial infarction or ischemia is not exclusionary.)
10. History of bleeding diathesis, hemorrhagic disorders, or coagulopathy; current use of anticoagulants or antiplatelet agents including warfarin, heparin, aspirin >325 mg/day, ticlopidine, clopidogrel, or cilostazol, unless discontinued ≥10 days prior to first dose and coagulation parameters meet inclusion criteria.
11. Severe infection requiring intravenous antibiotics, antifungals, or antivirals within 4 weeks prior to the first dose, or unexplained fever >38.5°C within 7 days prior to the first dose; baseline WBC >15 × 10⁹/L.
12. Known hypersensitivity to study drugs or excipients, or a history of severe hypersensitivity reactions such as generalized rash/erythema, hypotension, bronchospasm, angioedema, or anaphylaxis.
13. Conditions that may affect oral drug absorption, including dysphagia, nausea/vomiting, chronic diarrhea, or bowel obstruction.
14. Ongoing treatment with immunosuppressants or systemic corticosteroids (>10 mg/day prednisone or equivalent) within 2 weeks prior to the first dose.
15. Presence of any active autoimmune disease or a history of autoimmune diseases likely to recur (including but not limited to interstitial pneumonitis, uveitis, colitis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism). Exceptions include vitiligo and childhood asthma now in complete remission. Patients with asthma requiring bronchodilator therapy are excluded.
16. History of acute exacerbation of chronic obstructive pulmonary disease or other respiratory disease requiring hospitalization within 1 month prior to enrollment; patients with active tuberculosis or those who received anti-TB therapy within 1 year prior to screening.
17. HIV positive; or positive HBsAg with quantifiable HBV DNA ≥1000 cps/mL; or positive anti-HCV antibody.
18. Receipt of live vaccines within 4 weeks prior to first dose or anticipated during the study period.
19. Positive pregnancy test or currently breastfeeding.
20. Women of childbearing potential or sexually active men who are unwilling or unable to use medically accepted methods of contraception during the study period.
21. Any condition, as determined by the investigator, that may interfere with the study results or patient safety, such as substance abuse, serious physical or mental illness requiring concurrent treatment, significant laboratory abnormalities, or adverse social/family circumstances.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  Defined as the proportion of patients whose tumors shrink to complete response (CR) or partial response (PR) and remain for a certain period of time according to RECIST 1.1

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 1 year
  PFS is defined as the time interval from randomization to the observation of disease progression or death from any cause
Overall Survival (OS) | 1 year
  OS is defined as the time interval from randomization to death from any cause
Duration of Response (DOR) | 1 year
  DOR is defined as time from the first assessment of CR or PR until the date of the first occurrence of PD, or until the date of death
Disease Control Rate (DCR) | 1 year
  DCR is defined as the percentage of patients who have achieved CR, PR and SD to a therapeutic intervention
Adverse Events Reporting | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Health-related Quality of Life | 1 year
  Changes from baseline in patient-reported quality of life scores assessed every 2 cycles using the EORTC QLQ-C30 questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, version C30). The scores range from 0 to 100, with higher scores indicating a better quality of life outcome.
Head and Neck Cancer-Specific Quality of Life | 1year
  Changes from baseline in head and neck cancer-specific symptoms and functions assessed every 2 cycles using the EORTC QLQ-H&N35 module (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Head and Neck Cancer Module). The scores range from 0 to 100, with higher scores indicating a better quality of life outcome and lower scores indicating worse symptoms or functions.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Xiangya Hospital, Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No
Data can be requested from the corresponding author beginning 1 year after publication of the study.